CLINICAL TRIAL: NCT06108557
Title: A Prospective Study on the Role of Paraoxonase-1 Enzyme in Prediction the Severity and Outcome of Acute Organophosphate Poisoning and Its Correlation With Pseudo Cholinesterase Enzyme Level.
Brief Title: Paraoxonase-1 Pseudo Cholinesterase Organophosphate Toxicity Enzyme in Prediction the Severity and Outcome of Acute Organophosphate Poisoning and Its Correlation With Pseudo Cholinesterase Enzyme Level.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Abdelgawad, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-10-14MD
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Organophosphate Poisoning
MeSH Terms: conditions — Organophosphate Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Group I (Control group): which will include 20 healthy volunteers who will be selected based on their clinical examination, recent clinical history, and age and sex matching to the case group.This control group will be the basic profile for the studied group.
  Interventions: Diagnostic Test: Serum Pararoxonase -1 level; Diagnostic Test: Diagnostic Test: Serum pseudocholinesterase enzyme level
- case group (Active Comparator): Group II (Case group): which will include 70 cases, including both genders who will be admitted to Sohag University Hospital with acute organophosphate poisoning .
  Interventions: Diagnostic Test: Serum Pararoxonase -1 level; Diagnostic Test: Diagnostic Test: Serum pseudocholinesterase enzyme level

INTERVENTIONS:
Diagnostic Test: Serum Pararoxonase -1 level — The individual's venous blood will be taken five milliliters under strict aseptic conditions of both control and case groups (before antidotal therapy). Then the blood will be left to be coagulated for 10-20 minutes at room temperature, then centrifugation will be done by laboratory centrifuge. Serum samples were obtained, then half of the separated serum will be used for pseudocholinesterase enzyme assay and the other one will be used for Paraoxanase-1 (PON-1) analysis .
  Serum PON-1: The enzyme-linked immunosorbent assay (ELISA) will be used to measure it using human Pararoxonase (PON) ELISA kits.
  Serum pseudocholinesterase: is based on spectrophotometric measurement.
Diagnostic Test: Diagnostic Test: Serum pseudocholinesterase enzyme level — The individual's venous blood will be taken five milliliters under strict aseptic conditions of both control and case groups (before antidotal therapy). Then the blood will be left to be coagulated for 10-20 minutes at room temperature, then centrifugation will be done by laboratory centrifuge. Serum samples were obtained, then half of the separated serum will be used for pseudocholinesterase enzyme assay and the other one will be used for Paraoxanase-1 (PON-1) analysis .
  Serum PON-1: The enzyme-linked immunosorbent assay (ELISA) will be used to measure it using human Pararoxonase (PON) ELISA kits.
  Serum pseudocholinesterase: is based on spectrophotometric measurement.

SUMMARY:
The aim of the present study is to:

Evaluate the serum Paraoxonase-1 level in cases with organophosphate compounds poisoning and to correlate it᾿s level with the severity, outcome of acutely organophosphate poisoned cases .

Evaluate the serum pseudocholinestrase level in cases with organophosphate compounds poisoning and to correlate it with the Paraoxonase-1 level in those cases.

DETAILED DESCRIPTION:
Pesticides refer to a wide range of chemicals that are employed to increase agricultural output. Several pesticides have been shown to have severe negative impacts on human health, including acute toxicity (accidental poisoning deaths, particularly in impoverished nations) and chronic toxicity (even at low concentrations) (Trellu et al., 2021).

In the central nervous system of mammals and insects, organophosphate compounds (OPC) inhibit acetylcholinesterase irreversibly by inhibiting acetylcholine breakdown during nerve impulse transmission. Continuous neuronal excitation causes a variety of hazardous symptoms, including slow heart rate, pinpoint pupils, and seizures and respiratory failure (RF) which is the leading cause of morbidity and fatality (Zhai et al., 2021).

The diagnosis of acute organophosphate poisoning is based on the individual's medical history, physical examinations, and toxidromes of acute poisoning. Predicting the severity, prognosis, and complications related to poisoning requires a variety of clinical observations, electrocardiography, and blood or urine sample results. Electrolytes, the complete blood count, and arterial blood gas are virtually always tested (Kim et al., 2022).

Research started to focus on Paraoxonase-1 enzyme after terrorists released sarin in a Tokyo subway in 1995, which resulted in several deaths (La Du, 1996 ). Scientists searched for a potent enzyme for the rapid clearance of nerve agents (Josse et al., 2001).

Paraoxonase-1 (PON1) is an esterase that protects low-density lipoproteins from oxidation and detoxifies organophosphates and nerve agents. Paraoxonase-1 is predominantly produced in the liver, although enzyme activity has been detected in the kidney and brain (Schomaker et al., 2013).

They are found in a variety of tissues and are mostly linked to cell membranes and certain lipoproteins, while a free enzyme has been discovered in the blood (Reichert et al., 2021).

Initial baseline data suggests that Paraoxonase-1 varies among healthy people. Paraoxonase-1 exhibits broad range of specificity, affinity and different rates of hydrolysis for organophosphate compounds (Li et al., 2000).

Levels of plasma Paraoxonase-1 can vary tremendously, due to the polymorphisms in the promoter region of Paraoxonase-1 gene (Furlong, 2007).

Human serum Paraoxonase-1 hydrolyzes organophosphate compounds and so may significantly alters an individual᾿s susceptibility to the toxicity of these chemicals (Richard et al., 2013).

ELIGIBILITY:
Inclusion Criteria:

According to Patil (2014)'s recommendations, the following criteria are used to make the diagnosis of OPC poisoning:

Previous OPC exposure. The cholinergic toxidrome-specific features of OPC toxicity. After using atropine, muscarinic symptoms and signs improved. low pseudo-cholinesterase activity in serum.

Exclusion Criteria:

Cases under the age of 7. Asymptomatic cases. cases who have a history of severe renal, cardiac, pulmonary, or nephritic syndrome.

cases with any of the following conditions which reduce pseudocholinesterase activity: cases who have a history of parenchymal liver disease, acute infection, metastatic cancer, malnutrition, iron deficiency anemia, or dermatomyositis.

cases who are pregnant or who are using narcotics or poisonous substances (such as cocaine, carbon disulfide, benzalkonium salts, organic mercury compounds, ciguatoxins, and solanines) (oral contraceptive pills and metoclopramide).

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the serum Paraoxonase-1 level | 18 months
  Evaluate the serum Paraoxonase-1 level in cases with organophosphate compounds poisoning and to correlate it᾿s level with the severity, outcome of acutely organophosphate poisoned cases .
  the individual's venous blood will be taken five milliliters under strict aseptic conditions of both control and case groups (before antidotal therapy). Then the blood will be left to be coagulated for 10-20 minutes at room temperature, then centrifugation will be done by laboratory centrifuge. Serum samples were obtained, then half of the separated serum will be used for pseudocholinesterase enzyme assay and the other one will be used for Paraoxanase-1 (PON-1) analysis .
  Serum PON-1: The enzyme-linked immunosorbent assay (ELISA) will be used to measure it using human Pararoxonase (PON) ELISA kits.

SECONDARY OUTCOMES:
Evaluate Serum pseudocholinesterase level | 18 months
  Evaluate the serum pseudocholinestrase level in cases with organophosphate compounds poisoning and to correlate it with the Paraoxonase-1 level in those cases.
  Serum pseudocholinesterase: is based on spectrophotometric measurement.

REFERENCES:
- [Background] Furlong CE. Genetic variability in the cytochrome P450-paraoxonase 1 (PON1) pathway for detoxication of organophosphorus compounds. J Biochem Mol Toxicol. 2007;21(4):197-205. doi: 10.1002/jbt.20181. PMID 17936934
- [Background] Josse D, Lockridge O, Xie W, Bartels CF, Schopfer LM, Masson P. The active site of human paraoxonase (PON1). J Appl Toxicol. 2001 Dec;21 Suppl 1:S7-11. doi: 10.1002/jat.789. PMID 11920913
- [Background] Kim YO, Kim HI, Jung BK. Pattern of change of C-reactive protein levels and its clinical implication in patients with acute poisoning. SAGE Open Med. 2022 Jan 30;10:20503121211073227. doi: 10.1177/20503121211073227. eCollection 2022. PMID 35127097
- [Background] La Du BN. Structural and functional diversity of paraoxonases. Nat Med. 1996 Nov;2(11):1186-7. doi: 10.1038/nm1196-1186. No abstract available. PMID 8898738